CLINICAL TRIAL: NCT05782049
Title: Ultrasound Characteristics of the Salivary Glands in Patients With Rheumatoid Arthritis
Acronym: EchoPR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RBHP 2019 COUDERC
Record Dates: First submitted 2023-03-02; First posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-01

CONDITIONS: Rheumatoid Arthritis; Sjogren's Syndrome; Sicca, Asthenia, Polyalgia Syndrome (SAPS)
MeSH Terms: conditions — Arthritis, Rheumatoid; Sjogren's Syndrome; Asthenia

STUDY DESIGN:
Intervention Model Description: It's a cross-sectional case-control study. The study will include patients with rheumatoid arthritis compared to patients with Sjögren's syndrome or Sicca, Asthenia, Polyalgia syndrome (SAPS).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group of case patients (Other): 1. Patients with Rheumatoid Arthritis
  2. Patients with Sjögren's Syndrome
  Interventions: Other: Ultrasound of the salivary glands; Other: Measurement of salivary flow; Other: A Schirmer test
- Group of control patients (Other): Patients with Sicca, Asthenia, Polyalgia Syndrome (SAPS)
  Interventions: Other: Ultrasound of the salivary glands; Other: Measurement of salivary flow; Other: A Schirmer test

INTERVENTIONS:
Other: Ultrasound of the salivary glands — Salivary gland ultrasound is, a non-invasive, non-irradiating and easily accessible examination, offers promising results for the diagnosis of primary SS. It allows the identification of changes in the homogeneity of the echostructure of the main salivary glands in the parotid and submandibular region.The patient lies on the examination table with the head slightly turned to the side opposite the gland being examined. The examination will be done on the parotid and submandibular glands on both sides.The parotid glands will be measured in length and width.The surface of the gland will be calculated: (length x width)/2.The sub-maxillary glands will be measured in length and surface.
  The exam will be performed in 10 minutes.
Other: Measurement of salivary flow — Saliva flow measurement, which consists of measuring the quantity of saliva that the patient can emit in 15 minutes
Other: A Schirmer test — A strip of blotting paper graduated from five to five millimeters is placed in the eye for 5 minutes, avoiding any corneal contact.

SUMMARY:
The prevalence of Sjogren's syndrome (SS) in rheumatoid arthritis (RA) patients varies from 3.5 to 31%. Between 30% and 90% of patients with (RA) have dry eye and/or mouth syndrome. To date, no studies have assessed whether RA patients have echostructural changes in their salivary glands suggestive of SS and the factors associated with these changes.The aim of this study is to investigate if there are changes in the echostructure of the salivary glands of RA patients, especially in patients with dry syndrome.

DETAILED DESCRIPTION:
The EchoPR study is an exploratory pathophysiology, cross-sectional, case-control study.

The aim is to study the echo-structure of the salivary glands of patients with RA ( group of 70 patients), in comparison to patients with SS (suspected of strong alteration of the echo-structure)(group of 70 patients) and patients with sicca, asthenia, polyalgia syndrome (SAPS)(group of 70 patients).

After a standard consultation with the rheumatologist, patients in each group will have an salivary gland ultrasound to assess the homogeneity of the echostructure of the parotid and submandibular salivary glands. A salivary flow measurement for 15 minutes and a Schirmer test to determine tear secretion for 5 minutes are also performed. All of these tests are performed during a single visit, so the total study time for the patient is one hour. Patient recruitment is expected to last 1 year.

ELIGIBILITY:
Inclusion Criteria:

Patient, male or female, over 18 years of age, followed in the Rheumatology Department of the Clermont-Ferrand University Hospital, capable of giving informed consent to participate in the research.

* For RA subjects: Diagnosis of rheumatoid arthritis meeting the ACR/EULAR 2010 classification criteria.
* For SS subjects: Diagnosis of primary Sjögren's syndrome meeting the ACR/EULAR 2016 criteria.
* For SAPS subjects: Patients with dry syndrome not meeting the criteria for SS

Exclusion Criteria:

* Not covered by social security
* Minors or adults under the protection of the law or under the protection of justice.
* Pregnant or breastfeeding women
* Refusal to participate
* Interference with results or classification bias: secondary causes of dry syndrome: Previous radiotherapy of the face and neck, AIDS, Hepatitis C, Sarcoidosis, Amyloidosis, Hyper-IgG4 syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2025-02-02 (Estimated); Study Completion 2026-02-02 (Estimated)

PRIMARY OUTCOMES:
OMERACT (Outcome Measures in Rheumatology) B-mode ultrasound homogeneity score greater than or equal to 2 in at least one of the 4 salivary glands | 10 minutes
  The echostructure of the gland will be graded from 0 to 4 according to the OMERACT score :
  * 0: normal appearance
  * Grade 1: minimal inhomogeneity without hypoechoic/anechoic areas
  * Grade 2: moderate inhomogeneity with focal hypoechoic or anechoic areas
  * Grade 3 severe inhomogeneity with diffuse hypoechoic or anechoic areas of the whole gland or fibrous gland

SECONDARY OUTCOMES:
Color Doppler ultrasound vascularity score of OMERACT greater than or equal to 2 on at least one of the 4 salivary glands | 10 minutes
  For each patient, 4 grades will be obtained (1 per gland); the highest grade obtained and the sum of the 4 grades will be combined.
  A rating of the Doppler vascularization according to the OMERACT criteria will then be performed:
  * 0: no Doppler signal in the parenchyma of the gland
  * 1 : focal or scattered Doppler signal in the gland parenchyma
  * 2 : diffuse Doppler signal <50% of the gland parenchyma
  * 3 : diffuse Doppler signal >50 % of the gland parenchyma
Surface of the submandibular salivary glands | 2 minutes
  The surface of the gland will be calculated: (length x width)/2.
Length and width of the parotid glands | 2 minutes
  During the ultrasound, the examination will be done bilaterally on the parotid and submandibular glands in B mode with measurement of the dimensions of the glands (length and width in the longitudinal and axial plane for the parotids, longitudinal for the submandibular)
Length of the submandibular glands | 2 minutes
  During the ultrasound, the examination will be done bilaterally on the parotid and submandibular glands in B mode with measurement of the dimensions of the glands (length and width in the longitudinal and axial plane for the parotids, longitudinal for the submandibular)

CONTACTS AND LOCATIONS:
Overall Officials: Marion Couderc, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France